CLINICAL TRIAL: NCT04210037
Title: A Multi-Center, Phase Ib/II Study of Combination Treatment of APG-1252 With Paclitaxel in Patients With Relapsed/Refractory Small Cell Lung Cancer
Brief Title: Study of APG-1252 Plus Paclitaxel in Patients With Relapsed/Refractory Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Ascentage Pharma Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: APG1252SU101
Record Dates: First submitted 2019-12-20; First posted 2019-12-24 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — pelcitoclax; Paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Intervention Model Description: APG-1252 at the selected dose-level on days 1, 8 and 15 plus a fixed-dose of paclitaxel 80 mg/m˄2 on days 1 and 8 of a 21-day cycle. There will be three dose-levels of APG-1252 (-1, 80 mg; 1, 160 mg; 2, 240 mg).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- APG-1252 160 mg (Experimental): intravenous infusion over 30 minutes on days 1, 8 and 15
  Interventions: Drug: APG-1252; Drug: Paclitaxel
- APG-1252 240 mg (Experimental): intravenous infusion over 30 minutes on days 1, 8 and 15
  Interventions: Drug: APG-1252; Drug: Paclitaxel
- APG-1252 80 mg (Experimental): intravenous infusion over 30 minutes on days 1, 8 and 15
  Interventions: Drug: APG-1252; Drug: Paclitaxel

INTERVENTIONS:
Drug: APG-1252 — APG-1252 (Ascentage Pharma) is a highly potent Bcl-2 family protein inhibitor with high binding affinity for Bcl-2, Bcl-xL and Bcl-w. APG-1252 possesses strong antitumor activity as a single-agent against tumor cells addicted to Bcl-2/Bcl-xL, and exhibits a much broader antitumor activity when combined with chemotherapeutic agents.
Drug: Paclitaxel — 80 mg/m˄2 on days 1 and 8 of a 21-day cycle
  Other Names: Abraxane

SUMMARY:
This is a multi-center, open-label, phase Ib/II study of combination therapy with APG-1252 plus paclitaxel in patients with relapsed/refractory small-cell lung cancer(SCLC). The phase Ib portion will be done using time-to-event continual reassessment method (TITE-CRM) methodology to determine the maximum tolerated dose (MTD)/recommended phase 2 dose (RP2D) of APG-1252 with a fixed dose of paclitaxel. The phase II portion will utilize a Simon two-stage design to determine the efficacy of the combination therapy with response rate as the primary endpoint.

DETAILED DESCRIPTION:
Upon enrollment, patients will undergo a comprehensive history and physical exam, along with baseline laboratory assessment. Baseline CT imaging will be required within 4 weeks prior to study entry. Archival tissue is mandatory; a fresh biopsy of the primary tumor or a metastatic lesion prior to initiation of therapy is optional and post-treatment tumor biopsy is strongly encouraged.

In the phase Ib portion, eligible patients will receive APG-1252 at the assigned dose-level on days 1, 8 and 15 plus a fixed-dose of paclitaxel 80 mg/m˄2 on days 1 and 8 of a 21-day cycle. There will be three dose-levels of APG-1252 (-1, 80 mg; 1, 160 mg; 2, 240 mg) with the first patient starting at dose-level 1 and subsequent patients at dose-levels determined by the TITE-CRM methodology. There will be no intra-patient dose-escalation. Patients will be continuously assessed for adverse events, including DLTs which are defined in the protocol. Response assessment by CT imaging will occur every 2 cycles and treatment will continue until progression of disease, unacceptable toxicity, patient preference to stop treatment, withdrawal of consent, or administrative discontinuation.

In the phase II portion, eligible patients will receive APG-1252 at the RP2D determined in the phase Ib portion on days 1, 8 and 15 plus paclitaxel 80 mg/m˄2 on days 1 and 8 of a 21-day cycle. Response assessment by CT imaging will occur every 2 cycles and treatment will continue until progression of disease, unacceptable toxicity, patient preference to stop treatment, withdrawal of consent, or administrative discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed SCLC
* Progression of disease on or after initial treatment with platinum-based therapy with or without thoracic radiotherapy; patients may have also received prior immunotherapy or other chemotherapy agents, except for paclitaxel; there is no limit on the number of prior treatment regimens allowed
* Male or non-pregnant, non-lactating female patients
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Adequate hematologic function as indicated by:

  1. Platelet count ≥ 100,000/mm˄3 Note: Use of transfusions or thrombopoietic agents to achieve baseline platelet count criterion is prohibited.
  2. Hemoglobin ≥ 9.0 g/dL
  3. Absolute neutrophil count (ANC) ≥ 1000/µL Note: Use of growth-factors to maintain ANC criterion prior to enrollment is not permitted.
* Adequate renal and liver function as indicated by:

  1. Serum creatinine ≤ 1.5 × upper limit of normal (ULN); if serum creatinine is > 1.5 × ULN, creatinine clearance must be ≥ 50 mL/min
  2. Total bilirubin ≤ 1.5 × ULN; If patient has Gilbert's syndrome, may have bilirubin > 1.5 × ULN
  3. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × ULN; for patients with known liver metastases, AST and ALT may be ≤ 5 × ULN
  4. Coagulation: activated partial thromboplastin time (aPTT) and prothrombin time (PT) ≤ 1.2 × ULN
* Patients with previously treated, clinically controlled brain metastases are allowed. Clinically controlled is defined as surgical excision and/or radiation therapy followed by at least 14 days of stable neurologic function and no evidence of central nervous system (CNS) disease progression as determined by CT or MRI within 14 days prior to study enrollment. Continued use of corticosteroids is permissible.
* Willingness to use contraception by a method that is deemed effective by the investigator by both males and female patients of child bearing potential and their partners throughout the treatment period and for at least three months following the last dose of study drug (postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential).
* Able to understand and willing to sign a written informed consent form
* Able and willing to comply with study procedures and follow-up examination

Exclusion Criteria:

* Receiving concurrent anti-cancer therapy (chemotherapy, radiation therapy, surgery, immunotherapy, hormonal therapy, targeted therapy, biologic therapy) or any investigational therapy within 14 days prior to the first dose of treatment, with the exception of hormones for hypothyroidism, estrogen replacement therapy (ERT), anti-estrogen analogs, or agonists required to suppress serum testosterone levels
* Continuance of toxicities due to prior treatment that do not recover to < grade 2, except for clinically insignificant toxicities such as lymphopenia or alopecia
* Known bleeding diathesis/disorder
* Recent history of non-chemotherapy induced thrombocytopenia associated a major bleeding episode within 1 year prior to study entry
* Active immune thrombocytopenic purpura (ITP), active autoimmune hemolytic anemia (AIHA), or a history of being refractory to platelet transfusions, within 1 year prior to the first dose of study drug
* Serious gastrointestinal bleeding within 3 months of study entry
* Use of therapeutic doses of anti-coagulants is an exclusion, including anti-platelet agents. Use of low-dose anticoagulation medications to maintain the patency of a central intravenous catheter or aspirin (<100 mg) for cardiovascular protection are permitted.
* Failure to recover adequately from prior surgical procedures, as judged by the investigator. Patients who have had major surgery within 28 days from study entry, and patients who have had minor surgery within 14 days of study entry are excluded. (Minor surgery is invasive operative procedure involving resecting skin or mucus membranes and connective tissue. Major surgery is an invasive operative procedure involving more extensive resection, such as body cavity opening or organ resection.)
* Unstable angina, myocardial infarction, or a coronary revascularization procedure within 180 days of study entry
* Active symptomatic fungal, bacterial and/or viral infection including, but not limited to, active human immunodeficiency virus (HIV) or viral hepatitis (B or C); testing for hepatitis B and C is not required for study enrollment
* Uncontrolled concurrent illness that would limit compliance with the study requirements, including, but not limited to: serious uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness
* Prior treatment with a Bcl-2/Bcl-xL inhibitor
* Prior treatment with paclitaxel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Primary Toxicity Endpoint: dose-limiting toxicity (DLT) | 21 days
  DLT will be will be assessed via CTCAE version 5.0
Preliminary efficacy assessment | 12 months
  Partial or complete response according to RECIST v1.1 criteria measured at anytime with 12 months of start of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Yifan Zhai, MD, PhD, Study Chair — Ascentage Pharma Group Inc.
Locations (8):
- United States (6):
  - BRCR Medical Center, Plantation, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Virginia Cancer Specialists, Fairfax, Virginia
- Australia (2):
  - Westmead Hospital, Westmead, New South Wales
  - Flinders Medical Centre, Bedford Park, South Australia

IPD SHARING:
Plan to Share IPD: No